CLINICAL TRIAL: NCT06463054
Title: Testing an Intergenerational Model of Suicide Risk in Mother-child Dyads
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Oregon (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephanie Stepp, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY23070061; R01MH132543 (NIH)
Record Dates: First submitted 2024-05-23; First posted 2024-06-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dialectical Behavior Therapy Skills Group Training (Experimental): The investigators will employ Dialectical Behavior Therapy Skills Training in order to experimentally manipulate maternal emotion dysregulation, our targeted mechanism.
  Interventions: Behavioral: Dialectical Behavior Therapy Skills Group Training
- Safety Planning Intervention (Experimental): Safety Planning Intervention (SPI) or SPI only for 6 months, such that all mothers with history of suicidal behavior + ER difficulties will receive SPI.
  Interventions: Behavioral: Safety Planning Intervention

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy Skills Group Training — The investigators will employ Dialectical Behavior Therapy Skills Training in order to experimentally manipulate maternal emotion dysregulation, the targeted mechanism.
  Arms: Dialectical Behavior Therapy Skills Group Training
Behavioral: Safety Planning Intervention — Safety Planning Intervention (SPI) or SPI only for 6 months, such that all mothers with history of suicidal behavior + ER difficulties will receive SPI.
  Arms: Safety Planning Intervention

SUMMARY:
The investigators are interested in learning more about how the role of mothers' emotions has on the transmission of suicide risk to children. Eligible participants will be invited to participate in a baseline assessment, and 4 follow-up assessments in the next year. This research study is a randomized control trial. Participants that choose to enroll are randomly assigned, that is by chance (like by flipping a coin) to receive DBT Skills Training or treatment as usual (TAU). Participants may also be selected for DBT skills training, it which would occur once a week for 6 months.

DETAILED DESCRIPTION:
Suicide is now the 2nd leading cause of death among children ages 10-14 (CDC, 2022). This proposal responds to this public health crisis by testing an intergenerational mechanistic model of suicide risk in children while simultaneously testing a prevention and intervention approach that could be immediately useful. The investigators focus on children whose mothers have a history of suicidal behavior (intent, planning, attempt) as an especially vulnerable group with increased risk for an early and persistent course of suicidal thoughts and behaviors (STB). Theory and research point to emotion regulation (ER) as a potential intergenerational mechanism of suicide risk transmission from mother to child. Maternal ER affects child ER development via maternal emotion socialization, whereby maternal responses to child's emotions (validating/supportive vs. invalidating/unsupportive) shape how the child identifies, expresses, and modulates their emotions. The investigators theorize that maternal ER, a prerequisite for optimal maternal emotion socialization, serves as a clinically and etiologically significant pathway through which maternal history of suicidal behavior impacts the development of ER and emerging STB into adolescence. This proposal maximizes impact by leveraging a randomized controlled trial of Dialectical Behavior Therapy (DBT) Skills Training to improve maternal ER and testing a mechanistic model of suicide risk transmission from mothers to their children during a critical developmental juncture for the emergence and exacerbation of STB. Mothers will be randomized (1:1) to 6 months of either DBT Skills Training + Safety Planning Intervention (SPI) or SPI only. This design ensures all at-risk mothers receive SPI, an empirically supported intervention to enhance motivation, problem-solving, and mitigate suicide risk. The investigators hypothesize that mothers with a history of suicidal behavior and current ER difficulties who are randomly assigned to DBT Skills Training+SPI will experience improvements in ER compared to mothers assigned to SPI only. Furthermore, these improvements in maternal ER will predict meaningful decreases in child STB from late childhood into early adolescence through improved maternal emotion socialization and subsequent child ER development. The investigators will enroll 250 mother-child dyads with children ages 9-11 to retain a final sample of 225 dyads across two groups of mother-child dyads: (1) n=150 affected mothers (history of suicidal behavior + current ER difficulties) who will be randomly assigned to one of the two intervention conditions, and (2) n=75 nonaffected mothers (no history of suicidal behavior + no ER difficulties or psychiatric diagnosis since child's conception) to establish typical child ER development. Mother-child dyads will complete repeated multimodal assessments of ER, maternal emotion socialization, and STB over 24 months: baseline (intervention initiation), 3 months (intervention mid-point) 6 months (intervention termination), 12- and 24-months (post-intervention follow-up) when children will be ages 11-13, a high-risk time for STB. Findings from this study will identify intergenerational mechanisms of suicide risk and provide an intervention and prevention model for mitigating suicide risk in mother-child dyads.

ELIGIBILITY:
Inclusion Criteria:

* Biological mothers with legal custody of target child between 9-11
* Confirmed lifetime Biological mothers with legal custody of target child between 9-11
* Confirmed lifetime history of suicidal behavior for mothers of suicidal behavior for mothers

Exclusion Criteria:

* Any mothers and children with major medical illnesses that might be associated with organic personality changes or ER difficulties (e.g. Parkinson's Disease, seizure disorders)
* Cardiac nervous system abnormalities that would influence physiological readings
* Previous DBT (Dialectical Behavior Therapy) in the last six months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female mothers
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Child Suicidal Thoughts and Behaviors | Baseline, All Follow-up time points (3, 6, 12, and 24 months
  Suicidal thoughts and behaviors will be assessed by the Columbia Suicide Severity Rating Scale (C-SSRS).
  C-SSRS will be scored with these domains, higher scores indicate worse outcomes Suicidal Ideation (Highest Level Endorsed 1-5) Intensity of Ideation (2-25) Suicidal Behavior (present during time period) Y/N Medical Damage for Attempt (0-5) Potential Lethality (if medical damage = 0) (0-2)
Child Suicidal Thoughts and Behaviors | Baseline, All Follow-up time points (3, 6, 12, and 24 months
  Suicidal thoughts and behaviors will be assessed the Intensity of Suicide Ideation Scale (SIS; PhenX Toolkit).
  Intensity of Ideation Subscale The sum ranges from 2 to 25, with the higher number indicating more intense ideation.

SECONDARY OUTCOMES:
Child Mental Health Outcomes | Baseline, All Follow-up time points (3, 6, 12, and 24 months)
  Child mental health problems will assessed using the Youth Self-Report (YSR; child reports).
  Youth Self-Report (YSR) The YSR is a 112-item self-report scale that measures problem behaviors using a 3-point Likert scale (0 = not true, 2 = somewhat or sometimes true, or 3=very true or often true). Raw scores are converted into standard scores. A standard score of 50 is average for a child's age and gender, with a standard deviation of 10 points. Higher scores indicate more problems. Each score is interpreted based on the T-Score and Percentile Score: Scores below the 95th percentile (approximate t-scores of 65 and below) are considered in the normal range, scores between the 95th and 98th percentile (approximate t-scores of 65-70) are considered to be in the borderline clinical range, and scores above the 98th percentile (approximate t-scores of 70 and greater) are considered to be in the clinical range.
Child Mental Health Outcomes | Baseline, All Follow-up time points (3, 6, 12, and 24 months)
  Child mental health problems will assessed using Child Behavior Checklist (CBCL; mother reports).
  The Child Behavior Checklist (CBCL) consists of 113 items that measure problem behaviors, each rated on a 3-point Likert scale. Raw scores are converted into standard scores. A standard score of 50 is average for a child's age and gender, with a standard deviation of 10 points. Higher scores indicate more problems. Each score is interpreted based on the T-Score and Percentile Score: Scores below the 95th percentile (approximate t-scores of 65 and below) are considered in the normal range, scores between the 95th and 98th percentile (approximate t-scores of 65-70) are considered to be in the borderline clinical range, and scores above the 98th percentile (approximate t-scores of 70 and greater) are considered to be in the clinical range.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie D Step, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will archive data with the NIMH Data Archive (NDA) in two locations: (1) National Database for Clinical Trials Related to Mental Illness (NDCT), and (2) the Research Domain Criteria Database (RDoC db). Dr. Stepp will set up an NDA Account with access to NUID tool, and complete and submit an NDA Data Sharing Agreement for the project. The final dataset will cover clinical course and outcome data collected during the proposed project period. All data will be de-identified prior to submission to the NDCT and RDoCdb, and the team will obtain informed consent from participants to share their de-identified data. The investigators will fully comply with all NIH and IRB guidelines for data transfer, as well as federal regulations, including HIPAA.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after accomplishment of each primary aim or objective, or upon publication of the project's primary results.